CLINICAL TRIAL: NCT00358605
Title: A Randomized Study to Compare Oral Appliances to Standard CPAP Therapy in Patients With OSAHS, and to Assess Its Safety, Tolerability and Efficacy and Preference Over CPAP for Its Short-term Use.
Brief Title: The Use of Oral Appliances as an Adjunct to Continuous Positive Airway Pressure (CPAP) in the Treatment of Obstructive Sleep Apnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H05-70075
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Obstructive Sleep Apnoea
Keywords: OSAHS; Oral Appliance; Hypopnoea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The Klearway™ oral appliance — See Detailed Description.

SUMMARY:
This study will look at whether patients with OSAHS already successfully treated with nasal CPAP could successfully use an oral appliance as a short-term treatment alternative and whether patients who could use an oral appliance as an alternative would actually avail of its use, and to assess their preference in terms of treatment modality. The combination of therapies if tolerated, will allow greater flexibility of treatment and opportunity for ongoing compliance in circumstances where CPAP cannot be used.

DETAILED DESCRIPTION:
Each patient will undergo a detailed history and physical examination with particular attention to symptoms related to sleep disorders, cardiovascular disease, medications, motor vehicle accidents, occupation and change in symptoms. Weight, height and neck circumference will be measured and BMI calculated and compared to previous measurements recorded in the medical chart. The research question we are exploring is whether the oral appliance approach is better in terms of successful treatment, compliance with treatment, safety and quality of life when compared to the conventional CPAP therapy in OSAHS. It is a cross over design. Consecutive patients who

* meet the eligibility criteria
* agree to a trial of therapy with the oral appliance
* give informed consent will be recruited.

Inclusion criteria - stable on C-PAP for at least 3 months, and Previous diagnostic polysomnography within 2 years, and Pre-treatment AHI 10-30 ( mild-moderate sleep apnea), and Compliance > 4hrs per night, and Are willing and able to give informed consent

Exclusion Criteria - AHI >30, or Oxygen Saturation < 85% for > 10% of study time during previous diagnostic PSG, Or less than 8 teeth per jaw Or not enough teeth in good periodontal health to allow retention of the appliance, Operates heavy machinery or motor vehicle as part of job, or Clinical evidence of severe tempero-mandibular joint dysfunction, or Previous Motor Vehicle Crash assoc. with sleepiness, or Major cardiovascular morbidity, or Medically complicated or medically unstable. Thirty patients will be recruited over a period of 1 year. Prior to treatment baseline ESS and SAQLI will be recorded. Physical attributes will be recorded and if BMI and neck circumference are unchanged from pre-treatment records PSG will be deemed unnecessary at this point. Baseline RDI, and snoring index off treatment, will be recorded using portable snoresat monitoring.

All patients will visit the dental clinic for fitting and adjustment of the Klearway appliance. The appliance will be advanced under supervision of the clinic and patients will be assessed at intervals of 2-4 weeks. Titration will be assessed clinically based on patient sleepiness, snoring, comfort, and maximal jaw adjustment. Snoresat monitoring will be repeated while wearing the appliance in the optimal position to ensure adequate titration. Once titration has been completed the patient will be asked to wear the appliance exclusively for a period of at least 7 days. Full PSG will be recorded after 7 days while using the appliance. ESS will be measured at the time of PSG. Treatment efficacy at this point will determine safety to continue using the appliance. Treatment failure will be defined as an ESS >4 over baseline an AHI of >20 or > 50% of pre-treatment baseline.

Patients will be seen and reassessed and informed of sleep study results. Patients able to use the appliance safely will be asked to continue to use their OSA treatments individually and will be allowed to decide themselves which mode of therapy they will use each night. Patients will keep a daily diary recording use of treatment modality, length of time worn and also location (home, vacation etc). At the end of the study patients will be seen and diaries collected. Satisfaction levels will assessed and side effects recorded. Objective CPAP compliance will be analysed by downloading CPAP machines. Future treatment preference in terms of either treatment or a combination will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* stable on C-PAP for at least 3 months, and
* Previous diagnostic polysomnography ithin 2 years, and
* Pre-treatment AHI 10-30 ( mild-moderate sleep apnea), and
* Compliance > 4hrs per night, and
* are willing and able to give informed consent

Exclusion Criteria:

* AHI >30, or
* Oxygen Saturation < 85% for > 10% of study time during previous diagnostic PSG;
* Or less than 8 teeth per jaw;
* Or not enough teeth in good periodontal health to allow retention of the appliance;
* Clinical evidence of severe tempero-mandibular joint dysfunction;
* Operates heavy machinery or motor vehicle as part of job;
* previous Motor Vehicle Crash assoc. with sleepiness;
* or major cardiovascular morbidity;
* or medically complicated or medically unstable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
This study will compare apnea-hypopnea index (AHI) before and during oral appliance use.

SECONDARY OUTCOMES:
This study will compare Epworth Sleepiness Score, arousal index and sleep efficiency index between before and during oral appliance therapy.
It will compare the change in Sleep Apnea Quality of Life Index while on CPAP from baseline to while on Oral appliance.
Overall treatment compliance
Overall sleepiness score (subjective)

CONTACTS AND LOCATIONS:
Overall Officials: John Fleetham, MD, FCRC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Acute Sleep Disorder Program, UBC Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Almeida FR, Mulgrew A, Ayas N, Tsuda H, Lowe AA, Fox N, Harrison S, Fleetham JA. Mandibular advancement splint as short-term alternative treatment in patients with obstructive sleep apnea already effectively treated with continuous positive airway pressure. J Clin Sleep Med. 2013 Apr 15;9(4):319-24. doi: 10.5664/jcsm.2576. PMID 23585745
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/23585745